CLINICAL TRIAL: NCT04143919
Title: Heart Failure IDentification in a High Risk Cardiovascular OutpatiEnt Population (HIDE)
Acronym: HIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLCZ696DGT01
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiovascular risk factors; NT-proBNP; NYHA assessment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A recent Cochrane analysis reported a high burden of HF in Latin America (Ciapponi et al 2016), reporting an incidence of HF of 199 cases per 100 000 person-years. A cross-sectional study of 633 individuals aged ≥ 45 years, randomly selected and registered in a primary care program in Brazil (Jorge et al 2016) reported 36.6% of patients with Stage A HF, 42.7% with Stage B, and and 9.3% with symptomatic HF (Stage C). In real world settings primary care physician may attend to up to 40 patients per day, which rose to as many as 70 patients per day during high season demand, meaning in some circunstances physicians may only have up to 12 minutes per patient so patients with HF may go unnoticed. The aim of this study is to assess the practicality of an algorithm to identify new cases of HF Stage C in subjects who are at risk of CV disease in real world high-volume ambulatory primary care settings in Central America.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with CV risk factors (Experimental): Subjects with 2 or more CV risk factors will be identified. Cardiovascular risk factors include hypertension, dyslipidemia, obesity, vascular disease, diabetes mellitus, chronic kidney disease, arrhythmia requiring therapy, moderate to severe valvular disease, history of alcohol abuse, smoking, cancer chemotherapy, or thoracic radiotherapy, and abnormal findings in the most recent ECG or thoracic X-ray.
  Interventions: Diagnostic Test: NYHA assessment; Procedure: Serum NT-proBNP concentration; Diagnostic Test: Transthoracic Ecocardiogram

INTERVENTIONS:
Diagnostic Test: NYHA assessment — The New York Heart Association (NYHA) functional classification of HF
Procedure: Serum NT-proBNP concentration — Subjects with NYHA score ≥ II will undergo a rapid, on site serum NT-proBNP test on the same day of the visit. Roche CARDIAC proBNP+ test, using the Cobas h 232 device, is a quantitative immunological test for the determination of NT-proBNP in heparinized venous blood.
Diagnostic Test: Transthoracic Ecocardiogram — Subjects with a serum NT-proBNP result of ≥ 125 pg/mL at Visit 1 will be referred to a study cardiologist for a transthoracic echocardiogram to assess LVEF and relevant structural heart disease

SUMMARY:
This is a pilot, multicenter, real-world, single-visit, low risk, phase IV interventional study to efficiently identify new cases of heart failure (HF) Stage C in subjects who are at risk of cardiovascular (CV) disease in high-volume ambulatory primary care settings in 3 countries in Central America.

DETAILED DESCRIPTION:
Subjects with 2 or more CV risk factors will be identified and will undergo an NYHA score assessment. If the NYHA score is ≥ II, the serum NT-proBNP concentration will be determined on-site on the same day. If the serum NT proBNP concentration is ≥ 125 pg/mL, the subject will be referred to a country specific central echocardiography laboratory for a transthoracic echocardiogram to measure the left ventricular ejection fraction (LVEF) and relevant structural heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Male or female patients aged > 60 years at the time of informed consent
3. Presence of at least 2 or more of the following risk factors for HF (CV risk factors already diagnosed prior to study visit according to the usual medical practice criteria and listed in the medical chart):

   1. Hypertension
   2. Dyslipidemia
   3. Obesity
   4. Vascular disease, including coronary artery disease, cerebrovascular disease, and peripheral vascular disease
   5. Type 1 or 2 diabetes mellitus
   6. Chronic kidney disease
   7. Arrhythmia requiring therapy
   8. Moderate to severe valvular disease
   9. History of alcohol abuse,
   10. History of smoking,
   11. History of cancer chemotherapy, or

   i. History of thoracic radiotherapy l. Abnormal findings in the most recent ECG or m. Abnormal findings in the most recent thoracic X-ray
4. Attendance at a primary care consultation for reasons not related to HF

Exclusion Criteria:

1. Previous diagnosis of HF
2. Diagnosis of terminal cancer (malignant tumor that may cause the subject's death in a short period: days, weeks, or a few months)
3. Echocardiogram performed within the 12 months before the primary care consultation

Ages: 61 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Number of Cases of HF stage C | 5 months
  Proportion of subjects with HF Stage C among those with 2 or more CV risk factors

SECONDARY OUTCOMES:
Comparison of number of subjects diagnosed with HF stage C | 5 months
  Comparison of the number of subjects diagnosed with l HF Stage C versus the time matched historical proportion at the same study sites
Percentage of subjects with CV risk factos | 5 months
  Percentage of subjects with each listed CV risk factor among those with HF Stage C
Percentage of subjects with CV risk factors among participating countries | 5 months
  Percentage of subjects with each listed CV risk factor among participating countries
Ratio of subjects with each listed CV risk factor between subjects with and without HF Stage C | 5 months
  Ratio of presence versus absence of each listed CV risk factor between subjects with overall HF Stage C and without HF
Incidence of equality of HF Stage C among participating countries | 5 months
  Proportion and equality of proportions of HF Stage C subjects among participating countries
Mean NT-proBNP levels among subjects diagnosed with HF Stage C versus subjects with no HF | 5 months
  Comparison of the mean NT-proBNP (≥ 125 pg/mL) levels among subjects diagnosed with overall HF Stage C versus subjects with no HF

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceutical
Locations (3):
- Novartis Investigative Site, Santo Domingo, Dominican Republic
- Novartis Investigative Site, San Salvador, El Salvador
- Novartis Investigative Site, Guatemala City, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.